CLINICAL TRIAL: NCT04424537
Title: The Metabolic Response to Reduced Branched-chain Amino Acids in Humans 2
Brief Title: SOAR-2: Intervening in Obesity Through Reduction of Dietary Branched Chain Amino Acids
Acronym: SOAR-2
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to lack of funding
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019-0701; A534245 (Other: UW Madison); SMPH/MEDICINE/ENDOCRINOL (Other: UW Madison); Protocol Version 3/1/2021 (Other: UW Madison)
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Diabetes
Keywords: Calorie restriction
MeSH Terms: conditions — Obesity; Diabetes Mellitus | interventions — Diet; Diet, Protein-Restricted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): A control group will consume 2 meal replacement beverages(MRBs) made with whey protein
  The control diet group will be provided with a protein powder which will provide all Amino Acids. Diets will be provided in unmarked containers, to ensure subjects will be blinded to the dietary group assignment.
  No overall calorie reduction will be implemented for any group.
  All subjects will receive recipes developed by clinical nutritionist in the study team. Theses recipes will maximize palatability and match energy density across all diets and total protein content.
  The subjects will be able to use multiple different recipes over the course of the study to prevent taste fatigue and dropout. Each subject is anticipated to replace 2 meals per day with a beverage.
  Interventions: Dietary Supplement: Control diet
- Low protein(LP) diet (Active Comparator): This group will consume 2 meal replacement beverages(MRBs) containing low protein (goal to reduce total protein by 2/3rds).
  LP diet group will be provided with a protein powder which will provide all Amino Acids. Diets will be provided in unmarked containers, to ensure subjects will be blinded to the dietary group assignment.
  No overall calorie reduction will be implemented for any group.
  All subjects will receive recipes developed by clinical nutritionist in the study team. Theses recipes will maximize palatability and match energy density across all diets and total protein content.
  The subjects will be able to use multiple different recipes over the course of the study to prevent taste fatigue and dropout. Each subject is anticipated to replace 2 meals per day with a beverage.
  Interventions: Dietary Supplement: Low protein diet
- Low branched-chain amino acids (BCAA) (Experimental): The group on low-BCAA diet will consume 2 meal replacement beverages (MRBs) per day made with BCAD2 (branched chain amino acid) powder (lacking BCAAs).
  BCAD2 powder(Mead Johnson) is a fortified medical food powder that does not contain the BCAAs isoleucine, leucine, or valine, but provides all other essential and nonessential AAs, carbohydrates, fat, vitamins, and minerals.
  No overall calorie reduction will be implemented for any group.
  All subjects will receive recipes developed by clinical nutritionist in the study team. Theses recipes will maximize palatability and match energy density across all diets and total protein content.
  The subjects will be able to use multiple different recipes over the course of the study to prevent taste fatigue and dropout. Each subject is anticipated to replace 2 meals per day with a beverage.
  Interventions: Dietary Supplement: Low branched-chain amino acids(BCAA) diet

INTERVENTIONS:
Dietary Supplement: Control diet — Meal replacement beverages made with whey protein
  Arms: Control
Dietary Supplement: Low branched-chain amino acids(BCAA) diet — meal replacement beverages (MRBs) made with BCAD2 powder (lacking BCAAs).
  Arms: Low branched-chain amino acids (BCAA)
Dietary Supplement: Low protein diet — meal replacement beverages(MRBs) containing low protein
  Arms: Low protein(LP) diet

SUMMARY:
One of the primary risk factors for the development of diabetes is obesity. While even moderate weight loss achieved by dieting can lead to improvements in metabolic health, reduced-calorie diets are notoriously difficult to sustain. Over the past decade, a number of groups have shown that low protein diets are associated with metabolic health in both rodents and humans. In particular, specific building blocks of protein- the branched chain amino acids (BCAAs) leucine, isoleucine, and valine - are associated with insulin resistance and diabetes in humans. Blood levels of the BCAAs decrease in humans fed a low protein diet, and we recently showed that reducing either dietary BCAAs or protein rapidly restored normal body composition and insulin sensitivity to diet-induced obese mice without reducing calorie intake.

Current study will test the metabolic role of dietary BCAAs in humans by completing an adequately powered, randomized controlled study. A total of 132 subjects stratified by gender will be randomized to one of three groups: 1) Control; 2) Low Protein; 3) Low BCAA. Subjects in each group will replace two meals a day (and 2/3rds of their baseline dietary protein) with meal replacement beverages based on either complete protein powder or a BCAA-free medical food for two months. Primary outcomes will be weight and fasting blood glucose levels. A number of secondary outcomes will also be assessed and blood, adipose, and fecal samples will be collected for integrated transcriptional and metabolomic pathway analysis to identify and compare the metabolic pathways affected by low protein and low BCAA diets.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 28 - 40 (overweight to obese)
* Baseline protein intake within normal adult ranges (15.1%-20.8% of calories from protein)
* Able and willing to give written informed consent
* Stable weight (within 5 lbs. for at least 3 months)
* Not taking (or willing to cease taking) vitamin/mineral supplements, unless prescribed for a specific medical disorder
* Not planning to begin a new exercise or diet program

Exclusion Criteria:

* Use of prescription medications for diabetes or weight-loss
* Diabetes - fasting glucose level of greater than 125 mg/dL and/or hemoglobin A1C( HbA1c or A1C) above 6.4%
* Use of and unwillingness to discontinue weight loss beverage or meal plans (e.g. SlimFast or Jenny Craig)
* Low baseline albumin or pre-albumin levels (below normal reference range)
* Significant anemia (Hemoglobin < 11 g/dL)
* Known bleeding disorder or platelet dysfunction
* Participating in intensive exercise training program (high to moderate intensity exercise greater than 210 minutes per week) or planning to start new exercise program during study period.
* Significant co-morbidities (including kidney disease, liver disease, GI disease, cardiovascular disease, respiratory disease, malnutrition, substance abuse, psychiatric disease, or a diagnosed eating disorder).
* Planned smoking cessation or attempt at smoking cessation during study period
* Inability to tolerate meal replacement beverages due to palatability
* Bariatric surgery, gastric banding or liposuction
* Current or past (within 1 year) use of illicit drugs
* Use of and unwillingness to cease taking vitamin/mineral supplements and other over the counter supplements (e.g.,cinnamon, protein powders) that are known to affect weight and/or glucose tolerance, unless prescribed for a specific medical disorder
* Allergy to racemethionine
* Lactose intolerance
* Pregnancy or plans to conceive within 4 months of visit 1

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in weight | Baseline, 30 (±7)days, 60(-3 to +7)days, 134(+7) days
  Change in participant weight
Change in fasting blood glucose level | Baseline, 30 (±7)days, 60(-3 to +7)days, 134(+7) days
  Change in the participant's fasting blood glucose level

SECONDARY OUTCOMES:
Change in the body composition (adipose mass) as measured by DXA/BIS | Baseline, 60(-3 to +7)days
  Dual energy X-ray absorptiometry (DXA) is a standard technique for the determination of body composition. DXA results will be used to calculate fat and lean mass composition. Total body Bioelectrical Impedance Spectroscopy (BIS) is a minimal risk procedure which enhances DXA as it permits the determination of intracellular water.BIS is used to calculate fat and fat-free mass composition. A formula will be used to combine BIS fat-free mass composition and DXA lean mass composition corrected by limb length, which allows a surrogate measurement of muscle mass.
Change in Insulin sensitivity | Baseline, 30 (±7)days, 60(-3 to +7)days, 134(+7) days
  Insulin resistance will be measured by HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) method. Insulin resistance reveals the dynamics between the participant's baseline (fasting) blood sugar and the responsive insulin levels.
  HOMA-IR healthy range: 1.0 (0.5-1.4), less than 1.0 means participant is insulin-sensitive which is optimal, above 1.9 indicates early insulin resistance, above 2.9 indicates significant insulin resistance.
Change in Fibroblast growth factor 21 (FGF21) levels | Baseline, 30 (±7)days, 60(-3 to +7)days
  Fibroblast growth factor 21 (FGF21) is a hormone which regulate insulin signalling in response to nutritional status. Levels of FGF21 induced in response to low protein diet and fasting will be measured using enzyme-linked immunosorbent assay(ELISA) assay.
Change in Energy expenditure as measured by resting metabolic rate | Baseline, 60(-3 to +7)days
  Energy expenditure will be calculated from resting metabolic rate. Resting metabolic rate is the energy required by the body to perform the most basic functions when body is at rest.
Change in Muscle function as measured by jump maximal height | Baseline, 60(-3 to +7)days
  Jumping mechanography will be used to quantify muscle function. Jumping mechanography involves 3 supervised jumps on a force measurement platform. Analysis will be conducted on variables associated with the highest achieved jump height of the 3 trials.
  In Jumping mechanography, participants perform two-leg maximal countermovement jumps on a force plate (Leonardo, Novotec, Pforzheim, Germany). Maximal jump height(meter) will be calculated using Leonardo software.
Change in Muscle function as measured by jump velocity | Baseline, 60(-3 to +7)days
  Jumping mechanography will be used to quantify muscle function. Jumping mechanography involves 3 supervised jumps on a force measurement platform.Analysis will be conducted on variables associated with the highest achieved jump height of the 3 trials.
  In Jumping mechanography, participants perform two-leg maximal counter-movement jumps on a force plate (Leonardo, Novotec, Pforzheim, Germany). Jump velocity [meter/sec] will be calculated using Leonardo software.
Change in Muscle function as measured by relative power of jump | Baseline, 60(-3 to +7)days
  Jumping mechanography will be used to quantify muscle function. Jumping mechanography involves 3 supervised jumps on a force measurement platform.Analysis will be conducted on variables associated with the highest achieved jump height of the 3 trials.
  In Jumping mechanography, participants perform two-leg maximal countermovement jumps on a force plate (Leonardo, Novotec, Pforzheim, Germany). Relative power of jump [Watt/kg] will be calculated using Leonardo software.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn B Davis, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No